CLINICAL TRIAL: NCT00800852
Title: Increased Expression of Adiponectin Receptor 2 in the Mononuclear Cells in Children With Prader-Willi Syndrome
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Dong-Kyu Jin, Samsung Medical Center
Other Study IDs: 2008-10-040
Record Dates: First submitted 2008-11-30; First posted 2008-12-02 (Estimated); Last update posted 2008-12-02 (Estimated); Status verified 2008-11

CONDITIONS: Obesity; Prader-Willi Syndrome
Keywords: adiponectin; adiponectin receptor; Prader-Willi syndrome
MeSH Terms: conditions — Obesity; Prader-Willi Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The inflammatory process is involved in the pathogenesis of obesity. Prader-Willi syndrome (PWS) is a genetic model of syndromic obesity. Adiponectin is an adipokine with potent anti-inflammatory properties, and its effect is mediated through adiponectin receptors 1 (adipoR1) and 2 (adipoR2).

Objective of this study is to compare the expression of adipoR1, adipoR2, and adiponectin in peripheral blood mononuclear cells (PBMCs) in PWS children and obese control and to correlate receptor expression with insulin sensitivity and obesity-related parameters.

ELIGIBILITY:
Inclusion Criteria:

* children with Prader-willi syndrome
* children with simple obesity

Exclusion Criteria:

* subjects with diabetes mellitus (fasting plasma glucose > 126 mg/dL with a 2-h oral glucose tolerance test value of >200 mg/dl)

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Fourteen children with PWS and control subjects
Sampling Method: Probability Sample

CONTACTS AND LOCATIONS:
Overall Officials: Don-Kyu Jin, M.D., Principal Investigator — Samsung Medical Center, Sungkyunkwan Uiversity School of Medicine